CLINICAL TRIAL: NCT04187833
Title: Phase II Trial of Nivolumab in Combination With Talazoparib in Patients With Unresectable or Metastatic Melanoma and Mutations in BRCA or BRCA-ness Genes
Brief Title: Nivolumab in Combination With Talazoparib in Melanoma and Mutations in BRCA or BRCA-ness Genes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE2619
Record Dates: First submitted 2019-12-02; First posted 2019-12-05 (Actual); Results first posted 2025-01-14 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Metastatic or Unresectable Melanoma
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Nivolumab; talazoparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Nivolumab + Talazoparib (Experimental): Nivolumab 480mg intravenously every 4 weeks (28 days) + Talazoparib 1mg orally daily
  Interventions: Drug: Nivolumab; Drug: Talazoparib

INTERVENTIONS:
Drug: Nivolumab — 480mg intravenously every 4 weeks (28 days)
  Other Names: Opdivo
Drug: Talazoparib — 1mg orally daily
  Other Names: Talzenna

SUMMARY:
The purpose of this study is to evaluate how effective the study drugs, nivolumab (also known as Opdivo®) and talazoparib (also known as Talzenna®) are when given as a combination treatment for unresectable or metastatic melanoma. The study team wants to know the effectiveness of these drugs together in treating cancer than if each study drug was given by itself.

DETAILED DESCRIPTION:
This is a phase II, single arm, multi-institutional, open label trial in a sample size of 37 primary or recurrent, unresectable or metastatic melanoma patients progressed on prior checkpoint inhibitor therapy with germline or somatic mutations in BRCA1/2 or BRCA-ness.

The primary objective of this study is to estimate the clinical efficacy of nivolumab plus talazoparib in patients with unresectable or metastatic melanoma with BRCA1/2 or other DNA damage repair mutations (defined as BRCA-ness)

Secondary objectives and their endpoints include progression free survival (PFS) defined as time from first dose of treatment until disease progression, treatment related adverse events, anti-tumor activity , and immune-related progression free survival (irPFS).

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have a germline or somatic DNA damage repair mutation including any one of the following: BRCA1, BRCA2, ATM, CHEK1, CHEK2, PALB2, RAD50, RAD51, NBN, BLM, BRIP1, ATR, PARP1, MDC1, DSS1, ERCC3, MRE11, HDAC2, FANCA, MLH3, MLH1, EMSY, BAP1, LIG4, LIG3, PRKDC, XRCC6. The result may have been obtained from one of the following test providers: Myriad Genetics, Invitae, Ambry, Quest, Color Genomics, IMPACT, Foundation Medicine (tissue or ctDNA based), Guardant, or another CLIA approved tissue and/or serum based next generation sequencing-based assay.
* Subjects must have histologically or cytologically confirmed diagnosis of primary or recurrent metastatic melanoma.
* Subjects must have received prior checkpoint inhibitor therapy (defined as anti-CTLA4 or anti-PD-1 or combination anti-CTLA4/anti-PD-1), either for metastatic or unresectable disease or adjuvant therapy.
* ECOG Performance status ≤ 2.
* Subjects must have normal organ and marrow function as defined below:

  * Hemoglobin ≥ 9.0 g/dl
  * Absolute neutrophil count ≥ 1,500/mcL
  * Platelet count ≥ 90,000/mcL
  * Bilirubin ≤ 1.5 x ULN (except in subjects with Gilbert Syndrome, who can have a total bilirubin < 3.0mg/dL)
  * AST (SGOT) ≤ 3.0 X upper limit of normal
  * ALT (SGPT) ≤ 3.0 X upper limit of normal
  * Serum Creatinine Clearance ≥ 30mL/minute. See section 7.1 for talazoparib dose adjustment for renal impairment.
  * CrCl< 30mL/minute has not been studied in talazoparib.
* Measurable disease as defined by RECIST 1.1 criteria
* During screening, while taking study drug, and until 5 months after taking the final dose of study drug, women of childbearing potential (WOCBP) must practice one of the following methods of birth control:

  * Use double-barrier contraception method defined as male use of a condom and female use of a barrier method (e.g., contraceptive sponge, spermicidal jelly or cream, diaphragm [always use with spermicidal jelly/cream]).
  * Use of hormonal contraceptives (oral, parenteral, vaginal, or transdermal) for at least 3 months before the first study drug administration.
  * Use of an intrauterine device.
  * Have a male partner who has had a vasectomy (at least 6 months prior to study enrollment).
  * Or must abstain from sexual intercourse completely.
* During screening, while taking study drug, and until 7 months after taking the final dose of study drug, men who are sexually active with WOCBP must practice one of the following methods of birth control:

  * Have had a vasectomy (at least 6 months prior to study enrollment).
  * Use double-barrier contraception method defined as male use of a condom and female use of a barrier method (e.g., contraceptive sponge, spermicidal jelly or cream, diaphragm [always use with spermicidal jelly/cream]).
  * Partner use of an intrauterine device.
  * Partner use of hormonal contraceptives (oral, parenteral, vaginal, or transdermal) for at least 3 months before the first study drug administration.
  * Or must abstain from sexual intercourse completely
* Subjects must have the ability to understand and the willingness to sign a written informed consent document.
* Ability to swallow pills.

Exclusion Criteria:

* Prior treatment with a PARP inhibitor.
* Prior anti-cancer therapy for melanoma less than 14 days prior to first dose of study drug.
* Known symptomatic brain metastases requiring steroids. Patients with previously diagnosed brain metastases are eligible if they have completed their treatment and have recovered from the acute effects of radiation therapy or surgery prior to study enrollment, have discontinued corticosteroid treatment for these metastases for at least 4 weeks and are neurologically stable.
* Subjects with uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Known HIV or AIDS-related illness HIV-positive subjects on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with talazoparib. In addition, these subjects are at increased risk of lethal infections when treated with marrow suppressive therapy. Appropriate studies will be undertaken in subjects receiving combination antiretroviral therapy when indicated.
* Prior organ transplantation including allogeneic stem-cell transplantation.
* Poorly controlled or uncontrolled autoimmune disease that might deteriorate when receiving an immunostimulatory agent. Subjects with vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition or prior therapy requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll. Patients with endocrinopathies controlled on replacement drugs are eligible.
* Major surgery within 4 weeks prior to study enrollment.
* Current use of corticosteroids at the time of study enrollment, EXCEPT for the following:

  * a. Intranasal, inhaled, topical steroids, eye drops or local steroid injection (eg, intra-articular injection)
  * b. Systemic corticosteroids at physiologic doses ≤10 mg/day of prednisone or equivalent
  * c. Steroids as premedication for hypersensitivity reactions (eg, CT scan premedication)
* Diagnosis of Myelodysplastic Syndrome (MDS)
* Active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection at screening (positive HBV surface antigen or detectable HCV RNA if anti-HCV antibody screening test positive).
* Current or anticipated use of a P-glycoprotein (P-gp) inhibitor (amiodarone, carvedilol, clarithromycin, cobicistat, darunavir, dronedarone, erythromycin, indinavir, itraconazole, ketoconazole, lapatinib, lopinavir, propafenone, quinidine, ranolazine, ritonavir, saquinavir, telaprevir, tipranavir, valspodar, and verapamil), P-gp inducer (avasimibe, carbamazepine, phenytoin, rifampin, and St. John's wort), or inhibitor of breast cancer resistance protein (BCRP) (curcumin, cyclosporine, elacridar [GF120918], and eltrombopag).
* Inability to swallow capsules or known intolerance to talazoparib or its excipients.
* Pregnant women are excluded from this study because animal studies have demonstrated that nivolumab and talazoparib may cause fetal harm when administered to pregnant women. Breastfeeding women are excluded from this study because nivolumab and talazoparib may be excreted in human breastmilk and the potential for serious adverse reactions in nursing infants.
* Persisting toxicity related to prior therapy > Grade 1.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2020-06-05 (Actual); Primary Completion 2023-10-13 (Actual); Study Completion 2023-10-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Isaacs, MD, Principal Investigator — Cleveland Clinic Taussig Cancer institute, Case Comprehensive Cancer Center
Locations (1):
- Cleveland Clinic Taussig Cancer institute, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared to help protect the identity of our patients due to the small sample size and genetic information collected

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Nivolumab + Talazoparib
Started | 8
Completed | 7
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Nivolumab + Talazoparib
Number analyzed (Participants) | 8
Age, Customized [Count of Participants; unit: Participants]
  30-39 years old | 1
  40-49 years old | 1
  50-59 years old | 1
  60-69 years old | 3
  70-79 years old | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 8
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Best Overall Response as Defined by RECIST 1.1 Criteria
Description: Best overall response, defined as complete response (CR) and partial response (PR) by RECIST 1.1 criteria.
  Complete response (CR) is defined as the disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. Partial response (PR) is defined as a ≥30% decrease in the sum of the longest dimensions of the target lesions taking as a reference the baseline sum longest dimensions.
Time Frame: up to 24 months after treatment through study completion, an average of 2 years
Population: One patient out of 8 was enrolled but experienced a decline in health status before starting treatment and therefore did not receive any study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Nivolumab + Talazoparib
Number analyzed (Participants) | 7
Participants | 0

2. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS, defined as the time from the first dose of study treatment to the date of disease progression by RECIST 1.1 or death due to any cause, whichever occurs first.
  Progressive disease (PD) is defined as a ≥20% increase in the sum of the longest dimensions of the target lesions taking as a reference the smallest sum of the longest dimensions recorded since the treatment started, or the appearance of one or more new lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm.
Time Frame: up to 24 months after treatment through study completion, an average of 2 years
Measure: Median (Full Range); unit: Weeks
Arm/Group | Nivolumab + Talazoparib
Number analyzed (Participants) | 7
Weeks | 12 [6 to 24]

3. Secondary Outcome: Number of Participants With Treatment-related Adverse Events
Description: Number of participants with treatment-related adverse events, as assessed by National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) v5.0
Time Frame: 30 days after start of treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Nivolumab + Talazoparib
Number analyzed (Participants) | 7
Participants | 7

4. Secondary Outcome: Immune-related Overall Response (irOR) Defined by irRECIST
Description: Immune-related overall response (irOR), defined as immune-related complete response (irCR) and immune-related partial response (irPR) by irRECIST
Time Frame: up to 24 months after treatment through study completion, an average of 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Nivolumab + Talazoparib
Number analyzed (Participants) | 7
Participants | 0

5. Secondary Outcome: Immune-related Progression Free Survival (irPFS)
Description: irPFS, defined as the time from the first dose of study treatment to the date of disease progression by irRECIST
Time Frame: up to 24 months after treatment through study completion, an average of 2 years
Measure: Median (Full Range); unit: Weeks
Arm/Group | Nivolumab + Talazoparib
Number analyzed (Participants) | 7
Weeks | 12 [6 to 24]

6. Secondary Outcome: Overall Survival (OS)
Description: Overall survival (OS)
Time Frame: up to 24 months after treatment
Measure: Mean (Full Range); unit: Weeks
Arm/Group | Nivolumab + Talazoparib
Number analyzed (Participants) | 7
Weeks | 72 [21 to NA] — 1 participant still alive

7. Other Pre Specified Outcome: Anti-tumor Response as Measured by Immune-infiltration of Tumor Infiltrating Lymphocytes
Description: Anti-tumor response by measure of immune-infiltration of tumor infiltrating lymphocytes including flow cytometry on tumor biopsies and peripheral blood mononuclear cells (PBMCs)
Time Frame: At baseline, 12 weeks
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Patient Reported Outcomes for Adverse Events
Description: Patient reported outcomes for adverse events, as measured by PRO-CTCAE while on combination therapy
Time Frame: baseline and before each cycle (every 4 weeks) of nivolumab for a period of 12 months
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Evaluation of DNA Landscape as Described by Total Somatic Mutation Burden
Description: Evaluation of DNA landscape as described by total somatic mutation burden by DNA sequencing
Time Frame: At baseline, 12 weeks
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Gene Expression Analysis
Description: Gene expression by RNA sequencing
Time Frame: At baseline, 12 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: On or after Cycle 1 Day 1(each cycle is 28 days) through 30 days after the final dose of study drug, through study completion, an average of 3 years and 4 months
Description: All-cause Mortality: Only one death occurred within the study window due to disease progression and not related to toxicity from the treatment. The remaining deaths occurred after the study period had ended and were unrelated to the study treatment.
Arm/Group | Nivolumab + Talazoparib
All-Cause Mortality (participants affected / at risk) | 7/8
Serious Adverse Events (participants affected / at risk) | 1/8
Other Adverse Events (participants affected / at risk) | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nivolumab + Talazoparib (N=8)
Hepatobiliary disorders (Hepatobiliary disorders) | 1
Blood bilirubin Increased (Investigations) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nivolumab + Talazoparib (N=8)
Diarrhea (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 2
Dyspenea (Gastrointestinal disorders) | 2
vomiting (Gastrointestinal disorders) | 1
Belching (Gastrointestinal disorders) | 1
Abdominal Pain (Gastrointestinal disorders) | 1
Leukocytosis (Blood and lymphatic system disorders) | 1
Anemia (Blood and lymphatic system disorders) | 6
CPK decreased (Investigations) | 1
BUN decreased (Investigations) | 1
Paroxysmal atrial tachycardia (Cardiac disorders) | 1
Chills (General disorders) | 1
Edema Limbs (General disorders) | 1
Fatigue (General disorders) | 4
Non-cardiac chest pain (General disorders) | 1
Eye infection (Infections and infestations) | 1
Hepatitis viral (Infections and infestations) | 1
Fall (Injury, poisoning and procedural complications) | 1
White Blood Cells decreased (Investigations) | 4
Alanine aminotransferase increased (Investigations) | 1
Alkaline phosphatase increased (Investigations) | 2
Aspartate aminotransferase increased (Investigations) | 1
Blood bilirubin increased (Investigations) | 1
Blood lactate dehydrogenase increased (Investigations) | 1
CPK increased (Investigations) | 1
Weight loss (Investigations) | 1
Platelet count decreased (Investigations) | 1
CD4 lymphocytes decreased (Investigations) | 1
Anorexia (Metabolism and nutrition disorders) | 2
Hypercalcemia (Metabolism and nutrition disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 5
Hypernatremia (Metabolism and nutrition disorders) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 1
Hypocalcemia (Metabolism and nutrition disorders) | 1
Hypoglycemia (Metabolism and nutrition disorders) | 1
Hypolbuminemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 3
Arthralgias (Immune system disorders) | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 3
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2
Dizziness (Nervous system disorders) | 1
Depression (Psychiatric disorders) | 1
Anxiety (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 1
Confusion (Psychiatric disorders) | 1
Urinary Frequency (Renal and urinary disorders) | 1
Vaginal Discharge (Reproductive system and breast disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2
Pruritus (Skin and subcutaneous tissue disorders) | 1
Flushing (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-05-09): https://cdn.clinicaltrials.gov/large-docs/33/NCT04187833/Prot_SAP_000.pdf